CLINICAL TRIAL: NCT04281680
Title: Impact of Pasireotide on Postoperative Pancreatic Fistulas Following Distal Resections
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Tiina Vuorela, LL, attending surgeon, Helsinki University Central Hospital
Other Study IDs: Helsinki UCH
Record Dates: First submitted 2020-02-19; First posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Surgical Complications
MeSH Terms: interventions — pasireotide; Octreotide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pasireotide: Patients who received pasireotide perioperatively
  Interventions: Drug: Pasireotide 0.9 MG/ML
- Octreotide: Patients who received perioperative octreotide
- Control: Patients who received no additional medication in the timely cohort

INTERVENTIONS:
Drug: Pasireotide 0.9 MG/ML — 900-ug pasireotide administered subcutaneously twice daily for a week or until discharged from the hospital
  Other Names: Octreotide; Control, no-medication group
  Groups: Pasireotide

SUMMARY:
Between 2000 and 2016 258 distal pancreatectomies were performed at our University Hospital which were included in our analysis. Pasireotide was used in between July 2014 and April 2016. Patients received 900-ug pasireotide administered twice daily perioperatively. We analyzed patients who received octreotide treatment separately. Complications such as fistulas (POPF), delayed gas-tric emptying (DGE), postoperative hemorrhage (PPH), reoperations and mortality were recorded and analyzed 90 days postoperatively

DETAILED DESCRIPTION:
In total, between 2000 and 2016 in our University Hospital there were 276 elective distal pancreatectomies performed. In this retrospective cohort study, we included 258 of those distal pancreatectomy patients in the database in to our analysis. Pasireotide was administered preoperatively to all patients undergoing distal pancreatic resection between July 2014 to April 2016, as a part of a new practice in our clinic. One patient received both pasireotide and octreotide, for whom drug delivery was stopped after one day, and who was ex-cluded from analysis. We also excluded nine patients because insufficient data were found. Seven patients were excluded because they were recruited to another clinical study.

In total, 47 patients (18%) received 900-ug pasireotide administered subcutaneously twice daily for a week or until discharged from the hospital. We analyzed separately 31 (12%) patients who re-ceived octreotide peri-operatively. All other 180 (70%) distal resection patients operated on beween 2000 and 2016 constituted the control group.

The drug used in this study, pasireotide (Signifor), was supplied by Novartis Europharm Ltd. (Novartis, Basel, Switzerland). The drug manufacturer did not take part in the study nor did it cover any costs.

We collected information about the patient age, gender, the American Society of Anesthesiologists (ASA) Physical Status Classification, tumor histology and grade and type of resection. In addition, we recorded postoperative information, the length of the hospital stay, fever following surgery (>38 °C), complications and surgical and other re-operations.

ELIGIBILITY:
Inclusion Criteria:

All distal pancreatic resection patients in our time frame

Exclusion Criteria:

Included in another clinical trial, received both medications, inadequite patient records

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People who had pancreatic distal resection done between 2000 and 2016 at our institution.
Sampling Method: Non-Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
CR-POPF | 90 days
  clinically relevant postpancreatectomy fistula

SECONDARY OUTCOMES:
Postpancreatectomy complication | 90 days
  Any other surgical or no-surgical complication

IPD SHARING:
Plan to Share IPD: No
Data contains sensitive information, retrospective data analysis. no statements from participants to share information